CLINICAL TRIAL: NCT02937441
Title: Evaluation of the Cerebral Edema With Measurement of Optic Nerve Sheath in Children Having Diabetic Ketoacidosis
Brief Title: Evaluation of the Cerebral Edema in Children Having Diabetic Ketoacidosis
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ozlem Tolu Kendir, Fellow, Cukurova University
Other Study IDs: CUTF-GOKAEK-55-38
Record Dates: First submitted 2016-09-23; First posted 2016-10-18 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Edema
Keywords: C10.228.140.187
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Ultrasonic Measurement — How we measure;
  1. First measurement shall be taken in 4 hours.
  2. Second measurement shall be taken at 12 hours in mild and 12-18 hours measurement shall be taken for severe diabetic ketoacidosis,
  3. Third measurement shall be taken after fluid treatment.
  4. Fourth measurement shall be taken at patients polyclinic control.

SUMMARY:
The purpose of this study is to determine cerebral edema with evaluation of measurement of diameter of optic nerve sheath.

DETAILED DESCRIPTION:
The purpose of this study is to determine cerebral edema with evaluation of measurement of diameter of optic nerve sheath. For that, If patients have Fluid treatment shall be started in 4 hours in our or other Emergency Care, they will be included our study. If not, they will be out of our study.

How we measure;

1. First measurement shall be taken in 4 hours.
2. Second measurement shall be taken at 12 hours in mild and 12-18 hours measurement shall be taken for severe diabetic ketoacidosis,
3. Third measurement shall be taken after fluid treatment.
4. Fourth measurement shall be taken at polyclinic control. So, after all measurements will be hand and all data will be analyzed with statistical program. After that all outcome will be discussed and compared with patient at normal conditions at their polyclinic visit.

ELIGIBILITY:
Inclusion Criteria:

Fluid treatment shall be started in 4 hours in our or other Emergency Care

Exclusion Criteria:

Fluid treatment was started over four hours in other Emergency Care

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: General
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath diameters will be measured from 3 mm back of globe. | March 2017
  Optic Nerve Sheath diameters will be measured in Children Having Diabetic Ketoacidosis and compared with normal conditions at polyclinic.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem T Kendir, Dr. Fellow, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided